CLINICAL TRIAL: NCT07308808
Title: Intravesical Lactobacillus Crispatus: Clinical Safety and Microbiome Evaluation
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Medstar Health Research Institute (Other)
Collaborators: Loyola University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00008367; 7337853 (Other Grant/Funding Number: Craig H. Neilsen Foundation)
Record Dates: First submitted 2025-10-20; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Spinal Cord Injuries (SCI); Neurogenic Bladder; Urinary Tract Infection (Diagnosis)
MeSH Terms: conditions — Spinal Cord Injuries; Urinary Bladder, Neurogenic; Urinary Tract Infections; Disease | interventions — APF protein, Lactobacillus crispatus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Lactobacillus Crispatus bladder wash (Experimental): L. crispatus mixed with normal saline and instilled into the bladder will be used for intervention group. Subjects in the intervention group will be instructed to mix the contents of the applicator (by depressing the plunger, which extrudes the L. crispatus powder) into 45 cc of sterile 0.9% saline. After mixing, subjects will draw up the 45cc liquid L. crispatus mixture into a 60cc catheter tip syringe and instill via the intermittent catheter after the last catheterization prior to going to bed. Subjects will receive 2 doses (each in separate applicators) of L.crispatus and will repeat this process the following night 24 hours (+/- 2 hours) apart.
  Interventions: Drug: Lactobacillus Crispatus
- Saline Bladder Wash (Other): Subjects will draw up the 45cc sterile saline into a 60cc catheter tip syringe and instill via the intermittent catheter after the last catheterization prior to going to bed. Subjects will receive 2 doses of saline and will repeat this process the following night 24 hours (+/- 2 hours) apart.
  Interventions: Other: Saline bladder wash

INTERVENTIONS:
Drug: Lactobacillus Crispatus — L. crispatus mixed with normal saline and instilled into the bladder will be used for intervention group. Subjects in the intervention group will be instructed to mix the contents of the applicator (by depressing the plunger, which extrudes the L. crispatus powder) into 45 cc of sterile 0.9% saline. After mixing, subjects will draw up the 45cc liquid L. crispatus mixture into a 60cc catheter tip syringe and instill via the intermittent catheter after the last catheterization prior to going to bed. Subjects will receive 2 doses (each in separate applicators) of L.crispatus and will repeat this process the following night 24 hours (+/- 2 hours) apart.
  Arms: Lactobacillus Crispatus bladder wash
Other: Saline bladder wash — Subjects will draw up the 45cc sterile saline into a 60cc catheter tip syringe and instill via the intermittent catheter after the last catheterization prior to going to bed. Subjects will receive 2 doses of saline and will repeat this process the following night 24 hours (+/- 2 hours) apart.
  Arms: Saline Bladder Wash

SUMMARY:
The goal of this clinical trial is to determine whether Lactobacillus crispatus strains isolated from the lower urinary tracts of adult women can be used as an antibiotic-sparing treatment for urinary symptoms and urinary tract infection (UTI) among adults with neurogenic lower urinary tract dysfunction (NLUTD). The main question[s] it aims to answer are:

1. To identify soluble bactericidal compounds produced by urinary isolates of L. crispatus that kill uropathogenic E. coli (UPEC).
2. To determine if intravesical instillation of L. crispatus is safe and well tolerated in adults with NLUTD due to SCI who use intermittent catheterization (IC).

If there is a comparison group: Researchers will compare L. Crispatus to standard care saline to see if there is a difference in urinary symptoms and urinary microbiome.

Participants will be asked to complete daily symptom surveys, complete 2 bladder instillations, and collect, freeze, and return 14 urine samples.

DETAILED DESCRIPTION:
The investigators will conduct a 23-day pilot comparative study of L. crispatus instillation in 0.9% Sodium Chloride solution (saline) vs. saline solution only. Urine samples will be self-collected with a new or unused intermittent catheter and urinary symptoms will be monitored daily using the Urinary Symptom Questionnaire for Neurogenic Bladder-Intermittent Catheter (USQNB-IC). The investigators will obtain daily USQNB-IC electronically and urine samples for DNA sequencing for 7 consecutive days, and every 48 hours from days 11-23. The USQNB-IC will be completed on a daily basis until Day 23. On days 1-7, subjects will collect and freeze a daily urine sample (first urine of the day) in their home. On days 8 and 9, subjects will instill L. crispatus mixed in saline or saline solution only into their bladders immediately following the final catheterization of the day. Thus, each instillation will remain in the bladder overnight, and each instillation will occur ~24 hours (+/- 2 hours) apart. Starting on day 11, subjects will collect and freeze urine samples in their home every 48 hours, ending on day 23. Subjects will complete the USQNB-IC daily until day 23. At the end of the 23-day period, subjects will be given shipping materials including dry ice to assemble and overnight ship all the samples to Loyola University in Chicago, IL for processing, sequencing and analysis using FedEx at home pick-up. Staff at Loyola University Chicago are proficient and experienced in collecting and preparing urine samples for testing from research subjects. On Day 23, subjects will complete one final USQNB-IC and urine sample.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* SCI with at least 6-month duration
* NLUTD
* Utilizing intermittent catheterization for bladder management
* Community dwelling

Exclusion Criteria:

* Use of prophylactic antibiotics
* Instillation of intravesical antimicrobials to prevent UTI
* Psychological or psychiatric conditions influencing the ability to follow instructions
* Use of oral or IV antibiotics in the past 2 weeks
* Pregnancy
* Known genitourinary pathology beyond NLUTD
* Participation in another study that could confound results of the proposed study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-09-09 (Actual); Primary Completion 2027-03-30 (Estimated); Study Completion 2027-03-30 (Estimated)

PRIMARY OUTCOMES:
Urinary Symptom Questionnaire for Neurogenic Bladder-Intermittent Catheter | Daily for 23 days
  Will measure change in urinary symptoms for those that use an intermittent catheter. Higher scores may mean worse outcomes.
16S rRNA gene sequencing | days 1-7
  Changes in the presence and relative abundance of uropathogens and L. crispatus and saline solution
16S rRNA gene sequencing | alternating days 11-23
  Changes in the presence and relative abundance of uropathogens and L. crispatus and saline solution

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Groah, MD, Principal Investigator — MedStar National Rehabilitation Hospital
Locations (1):
- Medstar National Rehabilitation Hospital, Washington D.C., District of Columbia, United States